CLINICAL TRIAL: NCT02198391
Title: Multicenter Open-label, Randomized Clinical Trial to Assess the Safety and Efficacy of Echinaforce® Junior Tablets in Two Dosages for the Therapy of Common Cold Symptoms in Children (4-12 Years)
Brief Title: Study of Echinaforce Junior Tablets in Children With Acute Colds
Status: Completed | Type: Observational
Sponsor: A. Vogel AG (Industry)
Responsible Party: Sponsor
Other Study IDs: 920158
Record Dates: First submitted 2014-07-22; First posted 2014-07-23 (Estimated); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Respiratory Tract Diseases
MeSH Terms: conditions — Respiratory Tract Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 3 x 1 tablet per day: Echinaforce Junior tablets (low dose)
- 5 x 1 tablet per day: Echinaforce Junior tablets (high dose)

SUMMARY:
This study aims to investigate safety and efficacy of Echinaforce Junior tablets in two dosages of 3 x 1 and 5 x 1 tablets per day in children 4 - 12 years old with acute colds.

ELIGIBILITY:
Inclusion Criteria:

* age between 4 and 12 years
* signed informed consent by parents and optionally be the child
* daily access to computer / internet
* competence of german language

Exclusion Criteria:

* 13 years or older, younger than 4 years.
* presence of sinusitis, otitis media, pneumonia, bronchitis (complicated cold) at inclusion
* participation in a clinical study in the past 30 days
* intake of antimicrobial, antiviral, immunesuppressive substances, salicyl-containing medicines or bronchovaxom at first treatment period
* surgical intervention in the 3 months before inclusion or planned intervention during the observation period
* Known diabetes mellitus
* Known and treated allergic rhinitis, atopy or asthma
* cystic fibrosis, bronchopulmonic dysplasia, COPD
* immune system disorders, degenerative diseases (e.g. autoimmune disease like AIDS or leukosis)
* metabolic or resorptive disorders
* liver or kidney diseases
* serious health problems
* predisposition for complicated cold episodes in the judgement of the physician (sinusitis, otitis media, bronchitis, pneumonia)
* known allergy to plants of the compositae family (camomile or dandelion) or any of the substances of the investigational product

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children aged 4 - 12 years recruited in pediatrics practice
Sampling Method: Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2014-10-15 (Actual); Primary Completion 2015-08-07 (Actual); Study Completion 2015-08-07 (Actual)

PRIMARY OUTCOMES:
tolerability assessment by physicians | 4 months
  Within the observation period of 4 months a maximum of 3 colds can be treated with Echinaforce Junior tablets at the indicated dosage. At the exclusion visit the physicians rate the tolerability of Echinaforce Junior tablets as "very good", "good", "moderate" or "bad"

SECONDARY OUTCOMES:
tolerability assessment by parents/child | 4 months
  The tolerability of Echinaforce Junior is assessed after every acute treatment period of 10 days and after the observation period of 4 months
tolerability assessment by parents/child | 10 days
  The tolerability of Echinaforce Junior is assessed after every acute treatment period of 10 days and after the observation period of 4 months
Assessment of efficacy by parents/child | 4 months
  The acute efficacy of Echinaforce Junior is rated by the parents after every acute treatment period of 10 days as well as after the observation period of 4 months
Assessment of Cold Symptoms during Acute Treatment | 10 days
  During acute colds parents complete a symptom diary and assess cold-related symptoms (runny and congested nose, sneezing, headache, joint pain, sore-throat, fever, cough, shivering, sleep quality, additional care) in the child

CONTACTS AND LOCATIONS:
Overall Officials: Arnold Baechler, Dr. med., Principal Investigator — Facharzt FMH für Kinder- u. Jugendmedizin, Notkerstrasse 14 9006 St. Gallen, Switzerland
Locations (1):
- Dr. med. Arnold Bächler Facharzt FMH für Kinder- und Jugendmedizin, Sankt Gallen, Canton of St. Gallen, Switzerland